CLINICAL TRIAL: NCT00528229
Title: Multi-Slice CT of the Chest( MSCT Findings After Lung Transplantation)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Other Study IDs: KF 01 313267
Record Dates: First submitted 2007-09-11; First posted 2007-09-12 (Estimated); Last update posted 2007-09-12 (Estimated); Status verified 2007-06

CONDITIONS: CT of the Lung After Lungetransplantation

STUDY DESIGN:
Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Radiation: Computer Tomography

SUMMARY:
The purpose of the study is to compare Multi-Slice Computer Tomography findings with histological and physiological changes observed in transplanted lungs with Progressive Graft Disfunction.

ELIGIBILITY:
Inclusion Criteria:

* All patients that have had a lung transplantation

Exclusion Criteria:

* Under 18,
* Reduced kidney function,
* Known contrast allergy; and
* Language problems that make cooperation difficult.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2007-09

CONTACTS AND LOCATIONS:
Overall Officials: Esther Belmaati, MD, Principal Investigator — Department of Radiology, Rigshospitalet. Denmark
Locations (1):
- Department of Radiology, Rigshospitalet, Blegdamsvej 9, Copenhagen, Denmark